CLINICAL TRIAL: NCT02863666
Title: Verification of a Prediction Algorithm for Cardiopulmonary Patients Admitted to the Emergency Department (ED) (VPAC)
Brief Title: Verification of Prediction Algorithm
Acronym: VPAC
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 5703
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-12

CONDITIONS: Shortness of Breath Episode; Tachycardia; Bradycardia; Difficulty Breathing
Keywords: Cariopulmonary, cardiac arrest
MeSH Terms: conditions — Tachycardia; Bradycardia; Dyspnea; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective observational clinical study to verify an algorithm used to predict cardiopulmonary events in patients presenting to the emergency department.

DETAILED DESCRIPTION:
A novel algorithm for determining risk of acute cardiac complications, including cardiac arrest, for patients presenting to the ED has recently been reported. Unlike prior risk stratification tools that relied on basic vital sign data, this algorithm utilizes advanced computing of ECG data to solve the risk classification problem. Data will be collected on patients presenting to the emergency department with a primary complaint that is determined to be cardiopulmonary of origin by a clinician.

Verification of the results of the previous studies using this algorithm in a more diverse patient cohorts is required. As such, the proposed study will investigate the accuracy of the algorithm.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or older Admission to emergency department requiring immediate medical attention due to presumed cardiac or pulmonary cause(s) and considered 2nd or 3rd tier priority in triage system.

Exclusion Criteria:

Pregnant or suspected pregnancy Significant trauma Do Not Resuscitate order Known as Ward of the State

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting to the emergency department with cardiopulmonary related complaints
Sampling Method: Non-Probability Sample
Enrollment: 673 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurz, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - William Beaumont Hospital, Royal Oak, Michigan
- Antwerp University Hospital, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled: Enrolled subjects in observational study
Period: Overall Study
Arm/Group | Enrolled
Started | 673
Completed | 673
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled
Number analyzed (Participants) | 673
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304
  Male | 369
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 665
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 167
  White | 471
  More than one race | 0
  Unknown or Not Reported | 29
Region of Enrollment [Number; unit: participants]
  Belgium | 253
  United States | 420

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Cardiopulmonary Event
Description: The number of any cardiopulmonary event, not limited to:
  Cardiac arrest Sustained ventricular tachycardia (VT) Hypotension requiring inotropes or intra-aortic balloon pump (IABP) insertion Intubation or mechanical ventilation Complete heart block Bradycardia requiring insertion of a pacing wire or external pacing, and Percutaneous coronary intervention (PCI) or coronary artery bypass surgery (CABG)
Time Frame: Within 72 hours of presentation to ED
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 673
Participants | 145

2. Secondary Outcome: Cumulative Number of Cardiopulmonary Events in a Single Subject
Description: The cumulative number of any cardiac and cardiac-related events, not limited to:
  In-hospital Death In-hospital Cardiac Arrest Composite cardiovascular outcome or intervention (Lethal Arrhythmias , Acute Pulmonary Edema, Cardiogenic Shock, Myocardial Infarction, Percutaneous Coronary Intervention, Coronary artery Bypass Surgery , New or Recurrent MI, Recurrent Ischemia requiring Revascularization)
Time Frame: Within 72 hours of presentation to ED
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Arm/Group | Enrolled
All-Cause Mortality (participants affected / at risk) | 0/673
Serious Adverse Events (participants affected / at risk) | 0/673
Other Adverse Events (participants affected / at risk) | 5/673
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled (N=673)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT02863666/Prot_SAP_000.pdf